CLINICAL TRIAL: NCT01796860
Title: The Impact of Ankle Foot Orthosis (AFO) on Gait Recovery in Select Individuals With Multiple Sclerosis (MS)
Brief Title: Effectiveness of Ankle Foot Orthoses on Gait in Multiple Sclerosis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Modifications were made to protocol, new IRB pending
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Karen McCain, Assistant Professor, School of Health Professions, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MS AFO
Record Dates: First submitted 2013-02-18; First posted 2013-02-22 (Estimated); Results first posted 2015-08-03 (Estimated); Last update posted 2015-08-21 (Estimated); Status verified 2015-08

CONDITIONS: Multiple Sclerosis
Keywords: Gait; AFO; MS
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AFO (Other): All persons in the study will be fit with the same AFO (Tamarack joint with adjustable check strap).
  Interventions: Other: AFO

INTERVENTIONS:
Other: AFO — The purpose of this study is to investigate the impact of a specifically designed ankle foot orthosis (AFO, hinged, with tamarack joint and adjustable check strap) on the spatial and temporal gait parameters, electromyography (EMG), and walking endurance, in select individuals living with MS. Over the 13 week period, the subject will participate in 5 gait training sessions which will be at weeks 1, 2, 3, 7, and 10.

SUMMARY:
The purpose of this study is to investigate the impact of a specifically designed ankle foot orthosis (AFO, hinged, with tamarack joint and adjustable check strap) on the spatial and temporal gait parameters, electromyography (EMG), and walking endurance, in select individuals living with MS. This orthotic is fabricated to allow ankle range of motion required for normal gait kinematics. Additionally, it controls forward progression of the tibia during the stance phase of gait. This study has three hypotheses 1. Individuals who are fit with the AFO will demonstrate improvements in spatial and temporal gait parameters 2. Individuals who are fit with the AFO will demonstrate improvements in walking endurance, and 3. Individuals who are fit with the AFO will demonstrate improvements in muscle firing profiles/EMG measures.

DETAILED DESCRIPTION:
This is a non-randomized, single group (N=15), repeated measures study. The study will take place at the David M. Crowley Research and Rehabilitation Lab in the School of Health Professions at University of Texas Southwestern Medical Center. The outcome measures for the study include: 1. GAITRite System for temporal and spatial parameters, 2. EMG of the anterior tibialis, gastrocnemius, and vastus lateralis muscles, 3. 6 Minute Walk Test (gait endurance) 4. Lower extremity strength, 5. MS Fatigue scale, 6. Observational Gait Analysis - Video tape of over ground walking. This study will be 13 weeks long. Over the 13 week period, the subject will participate in 5 gait training sessions which will be at weeks 1, 2, 3, 7, and 10. They will be 60 minutes in duration. Outcome measures will be assessed at the following times: initial (T1), week 5 (T2), and week 13 (T3). Subjects will be closely monitored throughout the 13 week study and will be un-enrolled by self-request or the following medical reasons: 1. Acute exacerbation of MS symptoms, 2. New diagnosis with direct consequences affecting gait training, 3. Inability to tolerate the study AFO.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with a primary diagnosis of multiple sclerosis
* Individuals >21 and <60 years old
* Individuals who are able to maintain a walking velocity of 60 cm/sec for at least 2 minutes independently or with the use of a single tip assistive device.
* Current or past history of single or bilateral AFO use, including neuroprostheses
* Evidence of weakness in plantarflexors

Exclusion Criteria:

* The presence of co-morbidities (neuromuscular or musculoskeletal) that would negatively impact gait training
* Individuals with BMI with >/= 35kg/m2
* Individuals with range of motion deficit in the ankle limiting passive range of motion to neutral dorsiflexion
* Individuals that will begin the use of Ampyra during the course of the study
* Individuals for whom the cost of an orthosis would represent a financial burden
* Individuals who are receiving concurrent physical therapy services elsewhere,
* Multiple Sclerosis Neuropsychological Questionnaire (MSNQ) of >22
* Individuals for whom bilateral AFOs are indicated, but have different design

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2012-09; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen McCain, DPT, Principal Investigator — UTSW
Locations (1):
- University of Texas Southwestern Medical Center, School of Health Professions, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Ankle Foot Orthosis Group: All persons in the study will be fit with the same AFO (Tamarack joint with adjustable check strap).
  AFO: The purpose of this study is to investigate the impact of a specifically designed ankle foot orthosis (AFO, hinged, with tamarack joint and adjustable check strap) on the spatial and temporal gait parameters, electromyography (EMG), and walking endurance, in select individuals living with MS. Over the 13 week period, the subject will participate in 5 gait training sessions which will be at weeks 1, 2, 3, 7, and 10.
Period: Overall Study
Arm/Group | Ankle Foot Orthosis Group
Started | 10
Completed | 7
Not Completed | 3
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | Ankle Foot Orthosis Group
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.5 (5.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Change in Step Length From Initial Testing to End of Study
Description: Participants will be asked to walk on a 12-16 foot long vinyl pad placed on the floor. The mat will record and analyze step length.
Time Frame: Computerized gait analysis will be done at the time of enrollment and week 13.
Measure: Mean (Standard Deviation); unit: measure of length (cm)
Arm/Group | Ankle Foot Orthosis Group
Number analyzed (Participants) | 7
measure of length (cm) | 6.47 (3.26)

2. Secondary Outcome: Number of Participants With Change in Muscle Activity With Surface Electromyography (EMG) of Key Lower Extremity Muscles From Baseline to Final Testing
Description: Surface electromyography will be done on key muscles in the lower extremity (quadriceps, anterior tibialis, gastrocnemius) during computerized gait assessment. Changes in muscle activity would be things like large changes in amplitude of muscle firing or changes in the timing of muscle firing, for example. These would indicate changes in strength or perhaps motor learning as a result of wearing the ankle foot orthosis.
Time Frame: Surface EMG will be done at the time of enrollment and week 13.
Measure: Number; unit: participants
Arm/Group | Ankle Foot Orthosis Group
Number analyzed (Participants) | 7
participants | 0

3. Other Pre Specified Outcome: Change in Walking Endurance Using a 6-Minute Walk Test (6MWT) From Initial Testing to Final Testing
Description: Each participant will be asked to walk at a self-selected velocity on level surfaces for 6 minutes. They will be allowed to use assistive devices as necessary.
Time Frame: 6MWT will be done at the time of enrollment and week 13.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Ankle Foot Orthosis Group
Number analyzed (Participants) | 7
meters | 44.28 (77.12)

ADVERSE EVENTS:
Arm/Group | Ankle Foot Orthosis Group
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No